CLINICAL TRIAL: NCT04767347
Title: Renal Considerations in the Heat Stress Recommendations
Acronym: Aim1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Zachary J. Schlader, Associate Professor of Kinesiology, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1902420140
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Hot Weather; Adverse Effect; Kidney Dysfunction; Kidney Injury; Hyperthermia; Dehydration
MeSH Terms: conditions — Hyperthermia; Dehydration

STUDY DESIGN:
Intervention Model Description: This study will systematically examine the NIOSH recommendations for prescribing work-to-rest ratios during occupational heat stress on kidney function.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will not be directly informed of the experimental conditions and will be blinded to the hypotheses.
  The outcomes assessor will be blinded to the experimental conditions when analyzing the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed Work Rate (Experimental): Participants will walk on a treadmill at 3 mph and the grade will be adjusted to elicit 430 W of metabolic heat production (the most common work intensity). This study will systematically examine the NIOSH recommendations for prescribing work-to-rest ratios with increasing environmental heat stress (defined as Wet Bulb Globe Temperature, WBGT) at this fixed rate of metabolic heat production on kidney function.
  Interventions: Other: 23.0°C WBGT - Fixed Work Rate; Other: 25.5°C WBGT - Fixed Work Rate; Other: 27.5°C WBGT - Fixed Work Rate; Other: 28.5°C WBGT - Fixed Work Rate; Other: 35.5°C WBGT - Fixed Work Rate
- Fixed work-to-rest ratio (Experimental): This study will systematically examine the NIOSH recommendations on changes in kidney function when the work-to-rest ratio is fixed at 30 min per hour (the most commonly prescribed work-to-rest ratio), but the rate of metabolic heat production and environmental heat stress differs (Figure 2). As described in Study 1, the appropriate rate of metabolic heat production will be elicited by having participants walk on a treadmill at 3 mph and the grade will be adjusted accordingly.
  Interventions: Other: 26.0°C WBGT - Fixed work-to-rest ratio; Other: 30.5°C WBGT - Fixed work-to-rest ratio; Other: 30.5°C WBGT - Fixed work-to-rest ratio (high intensity)

INTERVENTIONS:
Other: 23.0°C WBGT - Fixed Work Rate — For four hours, participants will walk on a treadmill to elicit 430 W of metabolic heat production in the following conditions:
  23.0°C WBGT (29°C, 46% relative humidity) @ 60 min exercise per hour
  Arms: Fixed Work Rate
Other: 25.5°C WBGT - Fixed Work Rate — For four hours, participants will walk on a treadmill to elicit 430 W of metabolic heat production in the following conditions:
  25.5°C WBGT (31°C, 52% relative humidity) @ 45 min exercise per hour
  Arms: Fixed Work Rate
Other: 27.5°C WBGT - Fixed Work Rate — For four hours, participants will walk on a treadmill to elicit 430 W of metabolic heat production in the following conditions:
  27.5°C WBGT (33°C, 53% relative humidity) @ 30 min exercise per hour
  Arms: Fixed Work Rate
Other: 28.5°C WBGT - Fixed Work Rate — For four hours, participants will walk on a treadmill to elicit 430 W of metabolic heat production in the following conditions:
  28.5°C WBGT (34°C, 54% relative humidity) @ 15 min exercise per hour
  Arms: Fixed Work Rate
Other: 35.5°C WBGT - Fixed Work Rate — For four hours, participants will walk on a treadmill to elicit 430 W of metabolic heat production in the following conditions:
  35.5°C WBGT (40°C, 65% relative humidity) @ 15 min exercise per hour
  Arms: Fixed Work Rate
Other: 26.0°C WBGT - Fixed work-to-rest ratio — For four hours, participants will walk on a treadmill at differing levels of metabolic heat production and environmental conditions (noted below), but at a fixed work-rest ratio of 30 minutes per hour.
  26.0°C WBGT (31°C, 55% relative humidity) @ 530 W metabolic heat production
  Arms: Fixed work-to-rest ratio
Other: 30.5°C WBGT - Fixed work-to-rest ratio — For four hours, participants will walk on a treadmill at differing levels of metabolic heat production and environmental conditions (noted below), but at a fixed work-rest ratio of 30 minutes per hour.
  30.5°C WBGT (36°C, 55% relative humidity) @ 230 W metabolic heat production
  Arms: Fixed work-to-rest ratio
Other: 30.5°C WBGT - Fixed work-to-rest ratio (high intensity) — For four hours, participants will walk on a treadmill at differing levels of metabolic heat production and environmental conditions (noted below), but at a fixed work-rest ratio of 30 minutes per hour.
  30.5°C WBGT (36°C, 55% relative humidity) @ 530 W metabolic heat production
  Arms: Fixed work-to-rest ratio

SUMMARY:
An epidemic of chronic kidney disease is occurring in laborers who undertake physical work outdoors in hot conditions. The reason for this is unknown, but may be related to kidney dysfunction caused by increases in body temperature and dehydration. The current heat stress recommendations for workers were not developed with regards for kidney health. The purpose of this study is to determine if the current recommendations protect against kidney dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-44 y old
* Body mass index ≤35.0 kg/m2
* Self-reported to be healthy.

Exclusion Criteria:

* Not within defined age range
* Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2
* Deemed highly active according to the physical activity questionnaire (i.e., >3500 MET*min/wk)
* Body mass index >35.0 kg/m2
* Current or history of any renal disease, heart disease, stroke, immune or autoimmune disease, and/or gastrointestinal disease/surgery
* Hypertension during screening (systolic blood pressure >139 or diastolic blood pressure >89)
* Using medications that blunt the physiological response to exercise (e.g., beta blockers)
* Prescription medication with a known side effect of impaired temperature regulation or fluid balance (e.g., diuretics)
* Positive pregnancy test at any time during the study or breast feeding
* Current tobacco or electronic cigarette use or consistent use within the last 2 years
* Inability to safely complete the peak oxygen uptake test

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Peak urinary [IGFBP7•TIMP-2] | through study completion, up to 20 weeks
  Kidney injury marker

SECONDARY OUTCOMES:
Urinary NGAL | through study completion, up to 20 weeks
  Kidney injury marker
Urinary IGFBP7 | through study completion, up to 20 weeks
  Kidney injury marker
Urinary TIMP-2 | through study completion, up to 20 weeks
  Kidney injury marker
Urinary IL-18 | through study completion, up to 20 weeks
  Kidney injury marker
Urinary L-FABP | through study completion, up to 20 weeks
  Kidney injury marker
Renal artery blood velocity | through study completion, up to 20 weeks
  Index of kidney blood flow
Segmental artery blood velocity | through study completion, up to 20 weeks
  Index of kidney blood flow

OTHER OUTCOMES:
Core body temperature | through study completion, up to 20 weeks
  Heat strain variable
Mean skin temperature | through study completion, up to 20 weeks
  Heat strain variable
Oxygen uptake | through study completion, up to 20 weeks
  Heat strain variable
Heart rate | through study completion, up to 20 weeks
  Heat strain variable
Blood pressure | through study completion, up to 20 weeks
  Heat strain variable
Whole-body sweat rate | through study completion, up to 20 weeks
  Hydration and heat strain variable
Percentage change in body weight | through study completion, up to 20 weeks
  Hydration status variable
Plasma osmolality | through study completion, up to 20 weeks
  Hydration status variable
Urine osmolality | through study completion, up to 20 weeks
  Hydration status variable
Blood and plasma volume | through study completion, up to 20 weeks
  Hydration status variable
Urine specific gravity | through study completion, up to 20 weeks
  Hydration status variable
Plasma copeptin | through study completion, up to 20 weeks
  Hydration status variable
Creatinine clearance | through study completion, up to 20 weeks
  Kidney function variable
Fractional excretion of electrolytes | through study completion, up to 20 weeks
  Kidney function variable
Free water clearance | through study completion, up to 20 weeks
  Kidney function variable
Serum uric acid | through study completion, up to 20 weeks
  Kidney function variable
Urinary uric acid | through study completion, up to 20 weeks
  Kidney function variable

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health, Bloomington, Indiana, United States

REFERENCES:
- [Derived] Hess HW, Hite MJ, Heikkinen ME, Tarr ML, Tourula E, Johnson BD, Hostler D, Schlader ZJ. Critical Assessment of the Recommended Alert Limit Curves for Occupational Heat Exposure. Am J Ind Med. 2025 Nov;68(11):1004-1012. doi: 10.1002/ajim.70022. Epub 2025 Sep 7. PMID 40914830
- [Derived] Hess HW, Baker TB, Tarr ML, Zoh RS, Johnson BD, Hostler D, Schlader ZJ. Occupational Heat Stress Recommendation Compliance Attenuates AKI Risk Compared with a Work-Rest Ratio-Matched, Positive Control Scenario. Kidney360. 2023 Dec 1;4(12):1752-1756. doi: 10.34067/KID.0000000000000288. Epub 2023 Nov 1. PMID 37907448
- [Derived] Hess HW, Tarr ML, Baker TB, Hostler D, Schlader ZJ. Ad libitum drinking prevents dehydration during physical work in the heat when adhering to occupational heat stress recommendations. Temperature (Austin). 2022 Jul 20;9(3):292-302. doi: 10.1080/23328940.2022.2094160. eCollection 2022. PMID 36211944